CLINICAL TRIAL: NCT04901156
Title: A Randomized Pilot Trial of Repetitive Transcranial Magnetic Stimulation (rTMS) and Multi-Modality Aphasia Treatment (M-MAT) for Post-Stroke Non-Fluent Aphasia
Brief Title: rTMS and Multi-Modality Aphasia Therapy for Post-Stroke Aphasia
Acronym: TMAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Sean Dukelow, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB17-1014
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Stroke; Aphasia, Non-fluent
Keywords: Non-invasive brain stimulation; Transcranial Magnetic Stimulation; Multi-modality aphasia therapy; Neuroimaging; Stroke; Aphasia; Aphasia, Broca; Speech Disorders; Language Disorders
MeSH Terms: conditions — Stroke; Aphasia, Broca; Aphasia; Speech Disorders; Language Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-modality aphasia therapy plus 1Hz rTMS (Experimental): Chronic stroke patients, receive 10 days of 3.5hrs of multi-modality aphasia therapy (M-MAT) preceded by 20 minutes of 1Hz rTMS delivered at 100% of resting motor threshold over the right pars triangularis.
  Interventions: Device: 1Hz inhibitory rTMS; Behavioral: Multi-Modality Aphasia Therapy (M-MAT)
- Multi-modality aphasia therapy plus sham rTMS (Sham Comparator): Chronic stroke patients, receive 10 days of 3.5hrs of multi-modality aphasia therapy (M-MAT) preceded by 20 minutes of sham rTMS is achieved using a sham TMS coil which attenuates the magnetic output of the stimulator by 80%.
  Interventions: Behavioral: Multi-Modality Aphasia Therapy (M-MAT); Device: 1Hz sham rTMS

INTERVENTIONS:
Device: 1Hz inhibitory rTMS — 20 minutes of 1Hz (1200 pulses) repetitive transcranial magnetic stimulation (rTMS) applied by Magstim Rapid 2 stimulator equipped with an airfilm figure-8 coil
  Arms: Multi-modality aphasia therapy plus 1Hz rTMS
Behavioral: Multi-Modality Aphasia Therapy (M-MAT) — Participants receive 3.5 hours of intensive speech therapy in small groups delivered by a blinded speech language pathologist and therapy assistant. The objective of M-MAT is to improve word production through shaping of responses (ie. Gradually increasing complexity of spoken targets towards eventual mastery) and social-mediated repetitive practice. Therapists use game-based interactive tasks and rich multi-modal cueing (gestures, written words, drawing, reading words) to improve spoken production and oral communication.
Device: 1Hz sham rTMS — 20 minutes of 1Hz (1200 pulses) repetitive transcranial magnetic stimulation (rTMS) applied by Magstim Rapid 2 stimulator equipped with an airfilm figure-8 sham coil.
  Arms: Multi-modality aphasia therapy plus sham rTMS

SUMMARY:
Many stroke survivors experience aphasia, a loss or impairment of language affecting the production or understanding of speech. One common type of aphasia is known as non-fluent aphasia. Patients with non-fluent aphasia have difficulty formulating grammatical sentences, often producing short word fragments despite having a good understanding of what others are trying to communicate to them. Speech language pathologists (SLPs) play a central role rehabilitating persons with aphasia and administer therapy in an attempt to improve communication skills. Despite standard therapy, approximately 50% of individuals who experience aphasia acutely continue to have language deficits more than 6 months post-stroke.

In most people, Broca's area is dominant in the left side of the brain. Following a left-sided stroke, the right-sided homologue of Broca's area (the pars triangularis), may adopt language function. Unfortunately, reorganizing language to the right side of the brain seems to be less effective than restoring function to the left hemisphere. Repetitive transcranial magnetic stimulation (rTMS), a form of non-invasive brain stimulation, can be used to suppress activity of specific regions in the right side of the brain to promote recovery of function in the perilesional area. Despite preliminary success in existing studies using rTMS in post-stroke aphasia, there is much work to be done to better understand the mechanisms underlying recovery. Responses to rTMS have been positive, yet heterogenous, which may be related to timing of treatments following stroke.

ELIGIBILITY:
Inclusion Criteria:

* Isolated left middle cerebral artery (MCA) stroke more than 6 months ago (chronic)
* Stroke type: Ischemic or hemorrhagic
* Non-fluent aphasia as determined by the Western Aphasia Battery (Fluency < 5)
* Right-hand dominant prior to stroke
* English is first or primary language
* Ability to follow 3-step commands

Exclusion Criteria:

* Prior stroke to the right frontal lobe
* Current diagnosis of moderate to severe depression
* Diagnosis of any other psychiatric condition
* History of other neurologic disorders (e.g., epilepsy, brain tumor)
* Contraindication to MRI or TMS (metal in the head or any implanted electrical device)
* Has received intensive speech therapy within the past 6 months (>8 hours per week)
* Enrolled in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the Boston Naming Test within one week of intervention completion | Baseline, within 1 week of completing the 10 day intervention
  Number of spontaneously produced correct responses to a series of line drawings. That is, the number of correctly named images.
Change from baseline on the Boston Naming Test at 3 months | Baseline and 3-month follow-up
  Number of spontaneously produced correct responses to a series of line drawings. That is, the number of correctly named images.

SECONDARY OUTCOMES:
Trained and Untrained Picture Naming | Baseline, within 1 week of completing the 10 day intervention and 3-month follow-up
  Number of correctly named pictures from a set of trained nouns, trained verbs, untrained nouns, and untrained verbs
Story Narrative Task | Baseline, within 1 week of completing the 10 day intervention and 3-month follow-up
  Retelling of the Cinderella task as a measure of discourse, performance is quantified by number of correct information units.
Patient Health Questionnaire (PHQ-9) | Baseline, within 1 week of completing the 10 day intervention and 3-month follow-up
  A 9-item questionnaire completed by a caregiver to quickly assess depressive symptoms. The scale ranges from 0 to 27 with higher scores indicating greater endorsement of depressive symptoms.
EuroQoL-5D-5L | Baseline, within 1 week of completing the 10 day intervention and 3-month follow-up
  Assesses mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The answers given can be converted into EQ-5D index with scores anchored at 0 for death and 1 for perfect health. The EQ-5D also records the patient's self-rated health on a vertical visual analogue scale ranging from 0 to 100 with higher scores indicating higher self-perceived quality of life. This can be used as a quantitative measure of health outcome that reflects the patient's own judgement.

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available to other researchers

REFERENCES:
- [Result] Low TA, Lindland K, Kirton A, Carlson HL, Harris AD, Goodyear BG, Monchi O, Hill MD, Dukelow SP. Repetitive transcranial magnetic stimulation (rTMS) combined with multi-modality aphasia therapy for chronic post-stroke non-fluent aphasia: A pilot randomized sham-controlled trial. Brain Lang. 2023 Jan;236:105216. doi: 10.1016/j.bandl.2022.105216. Epub 2022 Dec 14. PMID 36525719